CLINICAL TRIAL: NCT06533046
Title: Ultrasound Estimation of Gastric Volumes in Patients With Previous Gastric Sleeve
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: 24-1278
Record Dates: First submitted 2024-07-23; First posted 2024-08-01 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-07

CONDITIONS: Aspiration
Keywords: gastric ultrasound; gastric sleeve procedure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to determine whether the existing model for calculating gastric volume based on an ultrasound-measured cross sectional area is accurate in adults who have had a previous gastric sleeve procedure. The main questions it aims to answer are:

Can the existing model accurately calculate gastric volume in patients who have had a previous gastric sleeve procedure?

If the existing model is not accurate in this population, can a model be developed to predict gastric volume in these patients based on ultrasound-measured cross section area?

Participants will be asked to fast prior to presenting for a gastric ultrasound scan. Following a fasted scan, patients will drink a small volume of water and undergo a second gastric scan.

DETAILED DESCRIPTION:
A major complication related to anesthesia in the perioperative period is aspiration of gastric contents. Multiple population level studies have found that aspiration among the leading causes of death from airway complications associated with anesthesia. In order to minimize the risk of aspiration, patients are often fasted prior to surgery if possible with the goal of emptying the stomach. Guidelines from the American Society of Anesthesiologists suggest that the existing evidence supports a 2 hour fast from clear fluids, a minimum of 6 hours from light foods such as toast, and even greater fasting times such as 8 hours or more from heavier foods such as meat. However, there is often a lack of clarity as to whether patients are adequately fasted prior to surgery especially elective surgery patients coming from home. This presents a dilemma of whether additional precautions need to be taken during surgery or even if the case needs to be cancelled.

One tool that has been used by anesthesiologists to clarify the risk of a full stomach preoperatively is an estimation of gastric volume using bedside ultrasound. The most commonly utilized method of estimating gastric volume is done by laying the patient in the right lateral decubitus position, measuring the diameter of stomach at the level of the antrum, and estimating a volume using the formula stomach volume (mL) = 27 + 14.6* antral cross sectional area (cm2) - 1.28*age (years). Volumes up to 1.5 mL/kg are generally thought to be consistent with baseline gastric secretions, while higher volumes or the presence of solids on ultrasound are indicative of a relatively full stomach and elevated aspiration risk. Gastric ultrasound and this method of estimating volume have been found to be very sensitive and specific for identifying a full stomach including in pregnant and severely obese patients.

Despite the proven accuracy of bedside ultrasound in estimating gastric volume in a variety of populations, all studies in the literature excluded patients who had previous gastric surgeries. There is a single published case study of an attempt to obtain an ultrasound estimate of gastric volume in a patient who had a previous roux-en-Y gastric bypass. This report found that the patient's stomach appeared to be empty on ultrasound regardless of ingested volume because the antrum of the stomach is no longer continuous with the remainder of the gastrointestinal tract after the operation. This is not the case in gastric sleeve procedures in which the greater curvature of the stomach is resected but the flow of material in the tract is left intact. Notably, an estimated 280,000 bariatric procedures were performed in the United States in 2022 with the vast majority of these being gastric sleeves. Given the large and ever increasing population of patients who have had gastric sleeve procedures and the proven utility of gastric ultrasound in assessing appropriate preoperative fasting it is important to determine whether traditional models of estimating gastric volume retain their accuracy in this population.

Participants will be asked to fast from solids for 8 hours and fluids for 2 hours prior to presenting for the study to ensure an empty stomach at baseline. They will be asked to lay on a flat surface on their right side. A curvilinear ultrasound probe will be placed on their abdomen and the antrum of the stomach will be identified with the liver and aorta in view at which point 3 measurements of both the anteroposterior and craniocaudal diameter of the stomach will be taken. These measurements will be used to calculate a gastric volume. Participants will then be asked to drink 100 mL of water. A second set of measurements of the gastric antrum will be obtained within 5 minutes of ingestion of the water as previously described. Serial measurements will be taken at thirty-minute intervals until 2 hours have past since ingestion. Participants will then be asked if they would be willing to repeat the above process at a later date. If they agree to go forward with an additional date, they will be asked to undergo the same process detailed above but with ingestion of 200 mL of water. If they are amenable to presenting a third time they will undergo a final trial with 300 mL of water as described above.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years of age
* English speaking
* Previous gastric sleeve procedure

Exclusion Criteria:

* Gastric surgery in addition to gastric sleeve
* Known hiatal hernia
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have previously undergone gastric sleeve procedure at UNC Hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2024-08-02 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Accuracy of existing gastric volume equation | 5 minutes after ingestion
  Calculated gastric volumes from after participants ingestion of a known quantity of water during the study will be compared to the known volumes of water that the subjects ingested using a mean squared error analysis.

SECONDARY OUTCOMES:
Equation for calculating gastric volume in patients with previous gastric sleeve | through study completion, an average of one year
  Should the existing model prove to be inaccurate, LASSO regression will be performed to identify a more accurate model in this population based on comparing the known volumes of water ingested and the measured cross sectional gastric area.
Gastric emptying time | 2 hours after ingestion
  The thirty-minute interval scans following ingestion will be used to determine the approximate time at which each patient is able to fully empty the volume of water they have ingested.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Doyal, MD, MPH, FASA, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available 9 to 36 months following publication and will be available indefinitely.
Access Criteria: The investigator who proposes to use the data must have approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and execute a data use/sharing agreement with UNC.

REFERENCES:
- [Background] Cook TM, Woodall N, Frerk C; Fourth National Audit Project. Major complications of airway management in the UK: results of the Fourth National Audit Project of the Royal College of Anaesthetists and the Difficult Airway Society. Part 1: anaesthesia. Br J Anaesth. 2011 May;106(5):617-31. doi: 10.1093/bja/aer058. Epub 2011 Mar 29. PMID 21447488
- [Background] Auroy Y, Benhamou D, Pequignot F, Bovet M, Jougla E, Lienhart A. Mortality related to anaesthesia in France: analysis of deaths related to airway complications. Anaesthesia. 2009 Apr;64(4):366-70. doi: 10.1111/j.1365-2044.2008.05792.x. PMID 19317699
- [Background] Practice Guidelines for Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration: Application to Healthy Patients Undergoing Elective Procedures: An Updated Report by the American Society of Anesthesiologists Task Force on Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration. Anesthesiology. 2017 Mar;126(3):376-393. doi: 10.1097/ALN.0000000000001452. No abstract available. PMID 28045707
- [Background] Perlas A, Mitsakakis N, Liu L, Cino M, Haldipur N, Davis L, Cubillos J, Chan V. Validation of a mathematical model for ultrasound assessment of gastric volume by gastroscopic examination. Anesth Analg. 2013 Feb;116(2):357-63. doi: 10.1213/ANE.0b013e318274fc19. Epub 2013 Jan 9. PMID 23302981
- [Background] Read MS, Vaughan RS. Allowing pre-operative patients to drink: effects on patients' safety and comfort of unlimited oral water until 2 hours before anaesthesia. Acta Anaesthesiol Scand. 1991 Oct;35(7):591-5. doi: 10.1111/j.1399-6576.1991.tb03354.x. PMID 1785235
- [Background] Phillips S, Hutchinson S, Davidson T. Preoperative drinking does not affect gastric contents. Br J Anaesth. 1993 Jan;70(1):6-9. doi: 10.1093/bja/70.1.6. PMID 8431336
- [Background] Harter RL, Kelly WB, Kramer MG, Perez CE, Dzwonczyk RR. A comparison of the volume and pH of gastric contents of obese and lean surgical patients. Anesth Analg. 1998 Jan;86(1):147-52. doi: 10.1097/00000539-199801000-00030. PMID 9428870
- [Background] Hausel J, Nygren J, Lagerkranser M, Hellstrom PM, Hammarqvist F, Almstrom C, Lindh A, Thorell A, Ljungqvist O. A carbohydrate-rich drink reduces preoperative discomfort in elective surgery patients. Anesth Analg. 2001 Nov;93(5):1344-50. doi: 10.1097/00000539-200111000-00063. PMID 11682427
- [Background] Kruisselbrink R, Gharapetian A, Chaparro LE, Ami N, Richler D, Chan VWS, Perlas A. Diagnostic Accuracy of Point-of-Care Gastric Ultrasound. Anesth Analg. 2019 Jan;128(1):89-95. doi: 10.1213/ANE.0000000000003372. PMID 29624530
- [Background] Kruisselbrink R, Arzola C, Jackson T, Okrainec A, Chan V, Perlas A. Ultrasound assessment of gastric volume in severely obese individuals: a validation study. Br J Anaesth. 2017 Jan;118(1):77-82. doi: 10.1093/bja/aew400. PMID 28039244
- [Background] Howle R, Sultan P, Shah R, Sceales P, Van de Putte P, Bampoe S. Gastric point-of-care ultrasound (PoCUS) during pregnancy and the postpartum period: a systematic review. Int J Obstet Anesth. 2020 Nov;44:24-32. doi: 10.1016/j.ijoa.2020.05.005. Epub 2020 May 29. PMID 32693329
- [Background] Pai SL, Bojaxhi E, Logvinov II, Porter SB, Feinglass NG, Robards CB, Torp KD. Ultrasound Assessment of Gastric Volume After Bariatric Surgery: A Case Report. A A Pract. 2019 Jan 1;12(1):1-4. doi: 10.1213/XAA.0000000000000824. PMID 29985844
- [Background] Clapp B, Ponce J, Corbett J, Ghanem OM, Kurian M, Rogers AM, Peterson RM, LaMasters T, English WJ. American Society for Metabolic and Bariatric Surgery 2022 estimate of metabolic and bariatric procedures performed in the United States. Surg Obes Relat Dis. 2024 May;20(5):425-431. doi: 10.1016/j.soard.2024.01.012. Epub 2024 Feb 1. PMID 38448343